CLINICAL TRIAL: NCT02584842
Title: Rivaroxaban for Thrombosis Prophylaxis in Endovenous Laser Ablation With and Without Miniphlebectomy: A Multicenter Experience
Brief Title: Rivaroxaban in Endovenous Laser Ablation With and Without Miniphlebectomy
Acronym: RITE
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2014-346
Record Dates: First submitted 2015-05-21; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Varicose Veins; Venous Thrombosis; Thromboembolism; Bleeding
MeSH Terms: conditions — Varicose Veins; Venous Thrombosis; Thromboembolism; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine retrospectively if the application of rivaroxaban after endovenous laser ablation with and without miniphlebectomy is safe and if it lowers the risk of venous thrombosis.

DETAILED DESCRIPTION:
Rivaroxaban is an orally active direct factor Xa inhibitor, that is used for thrombosis prophylaxis for example in the setting of orthopaedic surgery.

In the observed situation Rivaroxaban was applied in a dosage of 10mg daily during 5 days after endovenous laser ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients age greater than 18 years, informed consent was given.
* Endovenous Laser Ablation (EVLA) of the greater saphenous vein (GSV), autologous saphenous vein (ASV) and/or small saphenous vein (SSV) using 1470 nm wavelength radial laser (ELVeS, Biolitec, Austria) and postinterventional Endothermal Heat Induced Thrombosis (EHIT) prophylaxis with rivaroxaban.

Exclusion Criteria:

Patients are ineligible if they had:

* an endovenous ablation technique other than EVLA,
* other veins than GSV, ASV or SSV treated with EVLA (i.e. perforators),
* postinterventional EHIT prophylaxis other than prophylactic dose of rivaroxaban or
* informed consent was not given.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age greater than 18 years, informed consent was given. EVLA of the GSV, ASV and/or SSV using 1470 nm wavelength radial laser (ELVeS, Biolitec, Austria) and postinterventional EHIT prophylaxis with rivaroxaban.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with a EHIT class 3 or class 4 within 6 weeks after endovenous laser ablation | within 6 weeks after endovenous laser ablation

SECONDARY OUTCOMES:
Number of major or clinically relevant bleedings within 6 weeks after endovenous laser ablation. | within 6 weeks after endovenous laser ablation

CONTACTS AND LOCATIONS:
Overall Officials: Luca Spinedi, MD, Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Uthoff H, Holtz D, Broz P, Staub D, Spinedi L. Rivaroxaban for thrombosis prophylaxis in endovenous laser ablation with and without phlebectomy. J Vasc Surg Venous Lymphat Disord. 2017 Jul;5(4):515-523. doi: 10.1016/j.jvsv.2016.12.002. Epub 2017 Feb 21. PMID 28623988